CLINICAL TRIAL: NCT04790383
Title: Clinical Performance of Advanced Self-Adhesive Resin Composite Hybrid Restorations Versus Conventional Resin Composite Restorations in Posterior Teeth (1y Randomized Clinical Trial).
Brief Title: Clinical Performance of Advanced Self- Adhesivee Resin Composite Hybrid Restorations.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rawda Hesham Abd ElAziz (Other)
Responsible Party: Sponsor-Investigator, Rawda Hesham Abd ElAziz, lecturer at Conservative Dentistry department, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CU-2-2021
Record Dates: First submitted 2021-03-04; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Caries Class II; Caries,Dental
Keywords: self-Adhesive resin composite hybrid restorations; Posterior resin composite; Surefil One
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced Self-Adhesive resin composite hybrid restorations (Experimental): (Surefil one (Dentsply Sirona)).
  Interventions: Other: Advanced Self-Adhesive resin composite hybrid restorations (Surefil one (Dentsply Sirona)).
- Conventional resin composite restoration. (Active Comparator): Sphere Tec, (Dentsply Sirona)
  Interventions: Other: Conventional resin composite restoration. (Sphere Tec, (Dentsply Sirona

INTERVENTIONS:
Other: Advanced Self-Adhesive resin composite hybrid restorations (Surefil one (Dentsply Sirona)). — Hybrid resin composite that doesn't need bonding system and releases calcium and flouride.
  Arms: Advanced Self-Adhesive resin composite hybrid restorations
Other: Conventional resin composite restoration. (Sphere Tec, (Dentsply Sirona — Conventional Nanohybrid resin composite
  Arms: Conventional resin composite restoration.

SUMMARY:
Clinical performance according to modified USPHS criteria of advanced self-Adhesive resin composite hybrid restorations is evaluated for 1 year versus conventional resin composite restorations in posterior teeth.

ELIGIBILITY:
Inclusion Criteria:

* Patients with carious proximal cavities in molars
* Good oral hygiene.
* Presence of favorable occlusion and teeth are in normal contact with the adjacent teeth.

Exclusion Criteria:

* Teeth with signs and symptoms of irreversible pulpitis or pulp necrosis.
* Severe periodontal problems.

Ages: 17 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 63 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Clinical performance | Change from baseline at 6, 12 months
  Post operative Hypersensitivity, Secondary caries, Gross fracture, Cavo-surface marginal discoloration, Proximal contact.
  All these outcomes are measured by a score Alpha is excellent, Bravo is acceptable, Charlie is not accepted

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.dentsplysirona.com/en/explore/restorative/surefil-one.html